CLINICAL TRIAL: NCT00652574
Title: Phase I Trial of Induction Dasatinib Therapy in Patients With Resectable Malignant Pleural Mesothelioma
Brief Title: Dasatinib in Resectable Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0935; NCI-2010-01505 (Registry Identifier: NCI CTRP); W81XWH-07-1-0306 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2008-03-27; First posted 2008-04-03 (Estimated); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Malignant Pleural Mesothelioma; Dasatinib; BMS-354825; Sprycel; MPM
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dasatinib (Experimental): Dasatinib = BMS-354825, Sprycel
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — 70 mg by mouth twice daily x 28 days, for up to 2 years after surgery.
  Other Names: BMS-354825; Sprycel

SUMMARY:
The goal of this clinical research study is to learn how dasatinib affects biomarker levels in patients with malignant pleural mesothelioma that may be able to be removed by surgery. The safety and effectiveness of this drug will also be studied.

This research study is financially supported by the United States Department of Defense.

DETAILED DESCRIPTION:
The Study Drug Dasatinib is designed to decrease the activity of one or more proteins that are responsible for the uncontrolled growth of tumor cells. This may cause the tumor cells to die.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will take 2 dasatinib tablets by mouth 2 times a day for the 4 weeks before surgery (in the morning and 12 hours later). Dasatinib may be taken with or without food, but should be swallowed with at least 1 cup (8 ounces) of water. A light meal is not required, but may help you avoid getting a stomach ache when you take your dose. Tablets must be swallowed whole and may not be broken. If vomiting occurs within 30 minutes of swallowing the tablet(s), you can take another dose. If you miss a dose of dasatinib, take it as soon as you remember on the same day. If you miss taking your dose for 12 hours, take your regular dose the next scheduled day (do not take double your regular dose to make up for the missed dose). You will be given a "pill diary" to write down when you take the study drug. You will be shown how to fill it out and asked to bring the diary with you to each clinic visit.

Study Visits:

On Days 21 and 28, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of vital signs and weight.
* You will also have a test to check the amount of oxygen in your blood.
* Blood (about 3-4 teaspoons) will be drawn for routine tests.
* You will have a performance status evaluation.
* You will have an ECG.
* Blood (about 1-2 teaspoons) will be drawn to check your how well your blood clots.
* You will have a PET scan to check the status of the disease. This PET scan will be before your surgery, the study doctor will tell you when this will be performed.

Surgery:

After you have taken dasatinib for 28 days, you will have surgery to remove the tumor. You will continue to take the dasatinib until midnight the night before the surgery. Depending on the status of the disease, you will have either a pleurectomy or extrapleural pneumonectomy. You will be given a separate consent for these procedures, which will describe the surgery and any risks in detail.

Pleurectomy is the surgical procedure to remove the parietal pleura (the outermost lining around the lungs).

An extrapleural pneumonectomy is a surgical procedure that removes portions of the lung, the parietal pleura (the lining of the lung), the pericardium (the lining of the heart), and the diaphragm.

During surgery, 5-6 core biopsies, if possible, will be taken from different areas of the tumor for biomarker testing.

For the CT-guided core biopsy of the lung, a tissue sample is withdrawn from an organ or suspected tumor mass using a very thin needle and a syringe. The needle is guided while being viewed by the physician on a CT scan.

Length of Study:

After surgery, your doctor will decide the type of treatment you should receive for your condition. If the disease responded well to the 4 weeks of dasatinib, you may be eligible to continue taking dasatinib once a day starting 4-6 weeks after your surgery. The doctor may also decide that you can take dasatinib once a day starting 4-6 weeks after receiving radiation therapy. You may continue to take dasatinib as long as you are benefitting. You will be taken off study if intolerable side effects occur or the disease gets worse.

Follow-up Visits:

If you continue to receive the study drug after surgery, you will have a physical exam and a PET or CT scan every 8 weeks.

If you are taken off study for any reason, you will continue to be followed by the study team to see how you are doing.

This is an investigational study. Dasatinib is an investigational agent and ongoing clinical trials are using this drug in malignant mesothelioma. However, these studies have only recently started, and there is no information so far that shows the drug is effective in malignant mesothelioma. Dasatinib is FDA approved and commercially available for the treatment of acute lymphoid and chronic myeloid leukemia.

However, its use in this research study is investigational.

Up to 60 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with potentially resectable malignant pleural mesothelioma, IMIG stage I-III
2. Subject, age >/= 18 years
3. Any patient who is able to tolerate general anesthesia for the extended surgical staging and the definitive surgical resection.
4. No prior chemotherapy for mesothelioma within the last 3 years
5. No prior radiation to the area of primary disease. Radiation to chest wall port sites is acceptable.
6. No prior targeted biologic therapy (i.e. EGFR inhibitors, VEGF inhibitors) within the last 3 years
7. Adequate Organ Function: a) Total bilirubin < 2.0 times the institutional Upper Limit of Normal (ULN), b) Hepatic enzymes (AST, ALT ) </= 2.5 times the institutional ULN, c) Serum Na, K+, Mg2+, Phosphate and Ca2+>/= Lower Limit of Normal (LLN), d) Serum Creatinine < 1.5 time the institutional ULN, e) Hemoglobin, Neutrophil count, Platelets, PT, PTT all Grade 0-1
8. Ability to take oral medication (dasatinib must be swallowed whole)
9. Women of childbearing potential (WOCBP) must have: A negative serum or urine pregnancy test (sensitivity </= 25IU HCG/L) within 72 hours prior to the start of study drug administration
10. Persons of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 4 weeks after study drug is stopped
11. Signed written informed consent including HIPAA according to institutional guidelines

Exclusion Criteria:

1. Malignancy [other than the one treated in this study] which required radiotherapy or systemic treatment within the past 3 years.
2. Prior therapies to be excluded: any prior chemotherapy or targeted biologic therapy for mesothelioma used within the last 3 years
3. Concurrent medical condition which may increase the risk of toxicity, including: a) Clinically-significant coagulation or platelet function disorder (e.g. known von Willebrand's disease) b) Any disease which requires persistent anticoagulation therapy (and the patient may not be taken off the anti-coagulation safely) with coumadin, factor Xa inhibitors, or heparin (low-molecular weight, standard)
4. Cardiac Symptoms, consider the following: a) Uncontrolled angina, congestive heart failure or MI within (6 months), b) Diagnosed congenital long QT syndrome: 1. Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes), 2. Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec), 3. Subjects with hypokalemia or hypomagnesemia if it cannot be corrected
5. History of significant bleeding disorder unrelated to cancer, including: a) Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease), b) Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies), c) Ongoing or recent (</= 3 months) significant gastrointestinal bleeding
6. Concomitant Medications, consider the following prohibitions: a) Drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (Patients must discontinue drug 7 days prior to starting dasatinib): A) quinidine, procainamide, disopyramide, B) amiodarone, sotalol, ibutilide, dofetilide, C) erythromycin, clarithromycin, D) chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide E) cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine. F) moxifloxacin, levofloxacin
7. The concomitant use of H2 blockers or proton pump inhibitors with dasatinib is not recommended.The use of antacids should be considered in place of H2 blockers or proton pump inhibitors in patients receiving dasatinib therapy.a)Patient agrees to discontinue St. Johns Wort while receiving dasatinib therapy,b)Patient agrees that IV bisphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia,c)Patient may not be receiving any prohibited CYP3A4 inhibitors,d)Patient may not be receiving any alternative herbal remedies during the dasatinib treatment period
8. Women: a) are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after cessation of study drug, or, b) have a positive pregnancy test at baseline, or c) are pregnant or breastfeeding, d) Sexually active women of childbearing potential (WOCBP) must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized.,
9. -continued from exclusion #8-: e) Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy., f) All WOCBP MUST have a negative pregnancy test prior to first receiving dasatinib. If the pregnancy test is positive, the patient must not receive dasatinib and must not be enrolled in the study.
10. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-03-12 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Modulation of biomarker p-Src Tyr419 expression | Weekly during treatment followed by 5-6 core biopsies during surgery.
  McNemar's test used to compare the p-Src Tyr 419 expression before and after dasatinib treatment. The magnitude of modulation tested and quantified via paired-t test and Wilcoxon signed-rank test. For continuous data, paired-t test used for testing the biomarker modulation pre- and post-treatment.

SECONDARY OUTCOMES:
Progression-free Survival | 3 Years, or until disease progression.
  Kaplan-Meier method used to estimate the distribution of time-to-event-endpoints. Pearson and Spearman's correlation coefficients computed to correlate baseline biomarker values and biomarker modulation with participant's medical demographic variables as well as clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Anne S. Tsao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org